CLINICAL TRIAL: NCT06495723
Title: Phase I/II, Open-label, Multi-center Study to Evaluate the Safety and Efficacy of Glyco-humanized Polyclonal Antibody Directed Against Tumoral T Cells, in Patients With Relapsed/Refractory Peripheral T Cells Lymphoma (PTCL)
Brief Title: Polyspecific Antibodies in Lymphoproliferative T-cell Disorders
Acronym: PALT1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT 23-10; 2023-509648-88-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-18; First posted 2024-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Peripheral T Cells Lymphoma (PTCL)
Keywords: Relapsed Refractory PTCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation part: dose 2 mg/kg (Experimental): Dose Escalation part: Dose level of LIS1: 2 mg/kg.
  Interventions: Drug: LIS1
- Dose Escalation part: dose 4 mg/kg (Experimental): Dose Escalation part: Dose level of LIS1: 4 mg/kg.
  Interventions: Drug: LIS1
- Dose Escalation part: dose 6 mg/kg (Experimental): Dose Escalation part: Dose level of LIS1: 6 mg/kg.
  Interventions: Drug: LIS1
- Expansion part (Experimental): Expansion part: Participants will receive LIS1 at the RP2D determined in Part 1 of the study.
  Interventions: Drug: LIS1

INTERVENTIONS:
Drug: LIS1 — The study intervention (LIS1) is a glyco-humanized polyclonal antibody drug which is formulated for IV administration.

SUMMARY:
This is a 2-part study consisting of a Part 1, dose escalation and dose-finding component to establish the Maximal Tolerated Dose (MTD), or Recommended Part 2 Dose (RP2D) of LIS1 as a single agent; followed by a Part 2, to investigate anti-tumors efficacy of LIS1 in selected subtypes of Peripheral TCell Lymphoma (PTCL) and to further evaluate its safety and tolerability at RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed, written informed consent.
2. Is male or female, age ≥18 years old (at the time consent is obtained)
3. For Part 1: Has a histological diagnosis of the following relapsed or refractory PTCL based on WHO 2022 classification of lymphoid neoplasms

   * Intestinal T-cell and NK cell lymphoid proliferations and lymphomas (without NK cell neoplasms)
   * Hepatosplenic T-cell lymphoma
   * Anaplastic large cell lymphoma
   * Nodal TFH cell lymphoma
   * Other peripheral t-cell lymphomas For Part 2: The type of PTCL will be defined based on SC review after completion of Part 1 and will be documented in the protocol amendment
4. Had previously received 1 or more appropriate systemic therapies, including an alkylating agent and/or anthracycline, for treatment of the current disease (radiation therapy alone would not be acceptable as previous therapy). Participants with ALCL must have received prior brentuximab vedotin or be unable to receive it due to allergy or intolerance.
5. Experienced disease progression during or after completion of most recent therapy or refractory disease.
6. Has a measurable lesion by imaging: the longest diameter should be ≥1.5 cm for nodal lesions and >1 cm for extra-nodal lesions.
7. Experienced a toxicity of prior therapy: Participants must have recovered to less than Grade 1 or to baseline from toxicity of prior chemotherapy or biologic therapy and must not have had major surgery, chemotherapy, radiation, or biologic therapy within 2 weeks prior to beginning treatment.

   Note: Exceptions to this include events not considered to place the participant at unacceptable risk of participation in the opinion of the Investigator (e.g., alopecia).
8. Has either unstained tissues (block or unstained slides) or stained slides and pathology report available for central review. If stained slides or unstained tissue are not available or insufficient, a fresh tumor tissue sample is mandatory for central pathology. Central pathology confirmation is not required prior to enrollment.
9. Is able to provide a bone marrow aspirate and/or a biopsy no older than 3 months at screening and agrees to undergo post-treatment bone marrow aspirate or biopsy when required to confirm response.
10. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Has life expectancy of >3 months.
12. Has an adequate hematological and organ function at screening, including:

    * Hemoglobin ≥8.0 g/dL (prior transfusion is acceptable)
    * Absolute neutrophil count (ANC) ≥1000 cells/mm3 (without growth factor support within 7 days of ANC measurement)
    * Platelet count ≥50,000 cells/mm3 (without growth factor support or transfusion within 7 days of platelets measurement)
    * Creatinine clearance ≥30 mL/min
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × the upper limit of normal (ULN)
    * Serum total bilirubin <2 × ULN OR <3 × ULN (for participants with Gilbert's Syndrome)
13. Participants must be able to understand and sign an informed consent form.
14. All participants must use adequate contraception during participation in this study and for 6 months following completing therapy.

Exclusion Criteria:

1. Is diagnosed with a bulky disease (≥10 cm).
2. Has known history or presence of central nervous system involvement by leukemia or lymphoma.
3. Has Mature T-cell and NK-cell leukemias (WHO 2022 criteria)
4. Has T-lymphoblastic leukemia/lymphoma (WHO 2022 criteria)
5. Has tumor-like lesions with T-cell predominance (WHO 2022 criteria)
6. Has Primary cutaneous T-cell lymphomas (WHO 2022 criteria)
7. Has any other active cancers, or history of treatment for invasive cancer ≤3 years.

   Note: Participants with stage I cancer who have received definitive local treatment at least 3 years previously and are considered unlikely to recur are eligible. All participants with previously treated in situ carcinoma (i.e., non-invasive) are eligible.
8. Received any of the following treatments prior to the first dose of study medication:

   * Systemic chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks (or 5 half-lives, whichever is shorter) before Cycle 1 Day 1. Participants that received local radiation therapy are eligible.
   * Therapeutic anti-cancer antibodies <4 weeks
   * Any investigational drug in the last 4 weeks prior
   * Any major surgery or immunotherapy within 28 days
   * Toxin immunoconjugates <4 weeks
   * Nitrosoureas <6 weeks
   * Allogeneic hematologic stem cell transplant within 3 months
   * Adaptive cellular therapy such as autologous or donor natural killer cell or T lymphocyte infusions within 90 days
   * Systemic corticosteroids (prednisone or equivalent >10 mg daily) within 2 weeks prior to the start of therapy, or 12 weeks if given to treat graft versus host disease (GVHD), except for physiological replacement doses of cortisone acetate or equivalent
   * Systemic treatment for GVHD (including but not limited to oral or parenteral corticosteroids, ibrutinib, and extracorporeal phototherapy) within the last 12 weeks
9. Is experiencing a toxicity (or AE) from prior anti-cancer treatment that has not resolved to Grade ≤1 or baseline.
10. Has a known infection with human immunodeficiency virus (HIV) or serologic status reflecting active hepatitis B or C infection as follows:

    * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Participants with presence of HBcAb, but absence of HBsAg, are eligible only if hepatitis B virus (HBV) DNA is undetectable by an assay with sensitivity <20 IU/mL. If so, participants may either undergo regularly scheduled monitoring of HBV DNA or less frequent monitoring of HBV DNA while on prophylactic antiviral medication as defined by regional standard of care.
    * Presence of hepatitis C virus (HCV) antibody. Participants with presence of HCV antibody are eligible only if HCV RNA is undetectable.
11. Has a known active tuberculosis infection.
12. Has an active fungal, bacterial, and/or viral infection requiring systemic therapy.
13. Had a vaccination with a live vaccine within 35 days prior to the first dose of LIS1.
14. If woman, is pregnant or nursing a child.
15. Has an active autoimmune disease or history of autoimmune disease that may relapse except for type I diabetes under control, hypothyroidism managed with hormone replacement therapy, controlled celiac disease, and skin disease (vitiligo, psoriasis, etc.) not requiring systemic treatment.
16. Has a known history of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, acute lung disease, or dyspnea at rest or pulse oxymetrie < 92% at room air.
17. Has a clinically significant cardiovascular disease including the following:

    * Myocardial infarction or unstable angina within 3 months before screening
    * Congestive heart failure (New York Heart Association functional classification III-IV)
    * History of clinically significant arrythmias
    * QTcF > 470 msec
    * History of Mobitz II second degree or third-degree heart block without a permanent pacemaker in place
    * Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure >170 mm Hg and diastolic blood pressure >105 mmHg at screening
18. Has a cognitive impairment, active substance abuse, or psychiatric illness or social situations that, in the view of the Investigator, would preclude safe treatment or the ability to give informed consent and limit compliance with study requirements.
19. Has a known history of drug-induced liver injury, alcoholic liver disease, non- alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver or portal hypertension.
20. Has a hemophilia or von Willebrand's disease.
21. Has any psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
22. Has a concurrent condition that, in the Investigator's opinion, would jeopardize compliance with the protocol.
23. Are unable or unwilling to comply with study and/or follow-up procedures outlined in the protocol.
24. For France, participants under legal protection (safeguard, guardianship, curatorship).
25. Is currently participating in another therapeutic clinical study.
26. Has a known hypersensitivity to polyclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation part: Dose Limiting Toxicities (DLTs) | At the end of Cycle 1 (28 days)
  Incidence of DLTs in the first cycle
Dose Escalation part: treatment emergent adverse events (TEAEs) | After the first dose of study intervention through 60 days following the last dose of study intervention.
  The severity of averse events (AEs) will be graded according to the NCI CTCAE, v5.0.
  Treatment-emergent adverse events are defined as any AE with onset or worsening of a pre existing condition after the first dose of study intervention through 60 days following the last dose of study intervention.
Expansion part: Anti-tumors efficacy | Within 3 months after LIS1 initiation
  Objective response rate (ORR): defined as the proportion of participants with CR or PR assessed by Investigators according to Lugano criteria with the LYRIC modification for immunomodulatory drug.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of LIS: Cmax | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  LIS1 peak plasma concentration (Cmax) in plasma
Pharmacokinetics (PK) of LIS: Tmax | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Time to peak drug concentration in plasma (Tmax)
Pharmacokinetics (PK) of LIS: AUC | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  AUC24hours; AUC0-14days; AUC15-28days and AUC0-28days will be assessed
Pharmacokinetics (PK) of LIS: Ctrough | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Trough concentration (Ctrough) is the concentration reached by LIS1 immediately before the next dose is administered
Pharmacokinetics (PK) of LIS: Cmin | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Cmin for the minimum blood plasma concentration reached by LIS1 during the time interval between administration of two doses
Pharmacokinetics (PK) of LIS: T1/2 | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Half-life (T1/2) refers to the time required for plasma concentration of LIS1 to decrease
Pharmacokinetics (PK) of LIS: CL | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Clearance (CL) is the volume of blood or plasma cleared of LIS1 from the body per unit of time
Pharmacokinetics (PK) of LIS: Vd | At Cycle1Day 1 Predose and 5 minutes; 1; 2; 4; 8; 24 hours after the end of infusion. At Day1 and Day15 of Cycle2 to 6 (each cycle is 28 days): Predose and 5 minutes after the end of infusion. At Day 30 and Day60 after the last dose of LIS1.
  Volume of distribution (Vd) is defined as the total amount of LIS1 in the body divided by its concentration in plasma
Host immunogenicity to LIS1 | Before and after (up to 5 min after the infusion) LIS1 infusion at Cycle1Day 1, Cycle1Day8, Cycle1Day15, and Cycle1Day22, then before infusion at Day1 and Day15 of Cycle2 to Cycle6 (each cycle is 28 days), and at Day30 and Day60 after last dose of LIS1
  Number of participants who develop detectable anti-drug antibodies
Expansion part: treatment emergent adverse events (TEAEs) | After the first dose of study intervention through 60 days following the last dose of study intervention.
  The severity of averse events (AEs) will be graded according to the NCI CTCAE, v5.0.
  Treatment-emergent adverse events are defined as any AE with onset or worsening of a pre existing condition after the first dose of study intervention through 60 days following the last dose of study intervention.
Expansion part: Proportion of Complete Response (CR) as best overall response | Within 3 months and 6 months after LIS1 initiation
  Proportion of Complete Response as best overall response
Expansion part: Proportion of Partial Response (PR) as best overall response | Within 3 months and 6 months after LIS1 initiation
  Proportion of PR as best overall response
Expansion part: Proportion of Stable Disease (SD) as best overall response | Within 3 months and 6 months after LIS1 initiation
  Proportion of SD as best overall response
Expansion part: Proportion of Progressive Disease (PD) as best overall response | Within 3 months and 6 months after LIS1 initiation
  Proportion of PD as best overall response
Expansion part: Duration of response (DoR) | Within 3 months and 6 months after LIS1 initiation
  DoR: defined as the time interval between the first confirmed objective response (CR or PR) and the first occurrence of objective progression (PD) or death from any cause.
Expansion part: Time to response (TTR) | Within 3 months and 6 months after LIS1 initiation
  TTR: defined as the time from the date of LIS1 initiation to first confirmed objective response (CR or PR)
Expansion part: Progression-free survival (PFS) | Within 3 months and 6 months after LIS1 initiation
  PFS: defined as the time from the date of LIS1 initiation to the date of first documented progression or death
Expansion part: Overall survival (OS) | Within 3 months and 6 months after LIS1 initiation
  OS: defined as the time interval between the date of LIS1 initiation and the date of death due to any cause
Expansion part: Proportion of patients "bridged to transplantation" | Through study completion, an average of 1 year.
  Proportion of patients with a stem cell transplantation after LIS1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gandhi-Laurent DAMAJ, MD, Principal Investigator — University Hospital, Caen
Locations (8):
- France (5):
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Henri-Mondor, Créteil
  - CHU de Bordeaux - GH Sud - Hôpital Haut-Lévêque, Pessac
  - CHU de Lyon - Hôpital Lyon Sud, Pierre-Bénite
- Italy (3):
  - SC Ematologia Istituto Nazionale dei TumoriIRCCS Fondazione "G. Pascale", Napoli, Campania
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy